CLINICAL TRIAL: NCT01673789
Title: Phase 1/Phase 2 Study of Stem Cell Educator Therapy in Alopecia Areata
Brief Title: Stem Cell Educator Therapy in Alopecia Areata
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Collaborators: The First Hospital of Hebei Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-TH01
Record Dates: First submitted 2012-08-21; First posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Alopecia Areata
Keywords: Stem Cell Educator; Cord blood stem cells; Immune modulation; Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell Educator (Experimental): The collected lymphocytes are transferred into the device for exposure to CB-SCs, and other blood components are automatically returned to the patient. The Stem Cell Educator functions as part of a closed-loop system that circulates a patient's blood through a blood cell separator, briefly co-cultures the patient's lymphocytes with CB-SCs in vitro, and returns the educated lymphocytes to the patient's circulation. CB-SCs tightly attached to interior surfaces in the device, and only the CB-SC-educated autologous lymphocytes are returned to the subjects. The Stem Cell Educator therapy requires only two venipunctures with minimal pain, and does not introduce stem cells or reagents into patients.
  Interventions: Device: Stem Cell Educator

INTERVENTIONS:
Device: Stem Cell Educator — For the treatment, commonly the left (or right) median cubital vein, a patient's blood is passed through a Blood Cell Separator that isolates the lymphocytes from the blood according to the recommended protocol by manufacture; consequently, the collected lymphocytes were transferred into the Stem Cell Educator and treated by CB-SC; after that, the educated cells return the blood back to the patient via a dorsal vein of hand. During the MCS+ collection, the whole blood flow rate was maintained at 35 mL/min. The whole procedure was scheduled for 8 ~ 9 hrs.

SUMMARY:
Alopecia Areata (AA) is one of the most common T cell-mediated autoimmune diseases, leading to the chronic and relapsing hair loss. The prevalence of AA worldwide is 0.1 to 0.2%, affecting an estimated 5.3 million people in the United States. To date, the clinical therapies are limited and disappointed for the treatment of AA. Alternative approaches are needed. Increasing evidence demonstrates that stem cells possess the function of immune modulation. We established the Stem Cell Educator therapy by using cord blood-derived multipotent stem cells (CB-SCs)(Zhao Y, et al. BMC Medicine 2012). A closed-loop system that circulates a patient's blood through a blood cell separator, briefly co-cultures the patient's lymphocytes with adherent CB-SCs in vitro, and returns the educated lymphocytes (but not the CB-SCs) to the patient's circulation. Our clinical trial reveals that a single treatment with the Stem Cell Educator provides lasting reversal of autoimmunity that allows regeneration of islet beta cells and improvement of metabolic control in subjects with long-standing type 1 diabetes (T1D), which is another most common T cell-mediated autoimmune disorder in the United States. Here, we develop and explore the therapeutic effectiveness of Stem Cell Educator therapy in AA patients.

DETAILED DESCRIPTION:
A 16-gauge IV needle is placed in the left (or right) median cubital vein, and the patient's blood is passed through a Blood Cell Separator MCS+ (Haemonetics®, Braintree, MA) at 35 mL/min for 6 to 7 hours to isolate lymphocytes in accordance with the manufacturer's recommended protocol. The collected lymphocytes are transferred into the device for exposure to allogeneic CB-SCs (or process control without CB-SCs), and other blood components are returned to the patient. After 2 to 3 hours in the device, lymphocytes are returned to the patient's circulation via a dorsal vein in the hand under gravity flow control (2 to 3 mL/min) with physiological saline. Approximately 10,000 mL of blood is processed during the procedure resulting in approximately two repeated educations for the lymphocyte fraction. Patients are hospitalized for two days to monitor temperature and conduct routine laboratory blood tests for adverse reactions following treatment. Follow-up visits are scheduled 4, 12, 24, 40, and 54 weeks after treatment for clinical assessments and laboratory tests

ELIGIBILITY:
Inclusion Criteria:

* Patients are screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards recommended by the National Alopecia Areata Foundation (www.naaf.org).

Exclusion Criteria:

* Exclusion criteria are any clinically significant diseases in liver, kidney, and heart. Additional exclusion criteria are no pregnancy, no immunosuppressive medication, no viral diseases or diseases associated with immunodeficiency.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility and efficacy of Stem Cell Educator therapy in AA | 1 year
  The primary study end points are 1) feasibility of the Stem Cell Educator therapy in AA, 2) preliminary evaluation of the efficacy of the therapy for improving hire grow through a year.

SECONDARY OUTCOMES:
The efficacy of Stem Cell Educator therapy in modulating autoimmunity | 1 year
  The secondary study end point was evidence of the efficacy of the therapy in modulating autoimmunity. Baseline blood samples are collected prior to Stem Cell Educator therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhao, MD, PhD, Study Chair — Throne Biotechnologies Inc.
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Background] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Background] Zhao Y. Stem cell educator therapy and induction of immune balance. Curr Diab Rep. 2012 Oct;12(5):517-23. doi: 10.1007/s11892-012-0308-1. PMID 22833322
- [Derived] Li Y, Yan B, Wang H, Li H, Li Q, Zhao D, Chen Y, Zhang Y, Li W, Zhang J, Wang S, Shen J, Li Y, Guindi E, Zhao Y. Hair regrowth in alopecia areata patients following Stem Cell Educator therapy. BMC Med. 2015 Apr 20;13:87. doi: 10.1186/s12916-015-0331-6. PMID 25896390
- See also: Tianhe Stem Cell Biotechnologies Inc. — http://www.tianhecell.com